CLINICAL TRIAL: NCT04238208
Title: The Efficacy and Safety Profile of Capsaicin 8% Patch Versus 5% Lidocaine Patch in Patients With Diabetic Peripheral Neuropathic Pain: a Randomized, Placebo-controlled Study of South Asian Male Patients
Brief Title: The Efficacy and Safety Profile of Capsaicin 8% Patch Versus 5% Lidocaine Patch in Males With Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Dr Zainab Khan, Consultant, Endocrinology Unit, Department of Internal Medicine., Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LIDCAI38920
Record Dates: First submitted 2020-01-19; First posted 2020-01-23 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Nerve Problems; Diabetic Neuropathy; Diabetic Complications Neurological
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Lidocaine; Transdermal Patch; Capsaicin

STUDY DESIGN:
Intervention Model Description: This present study was a double blinded, placebo controlled, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study, the investigators, patients and care providers were not aware of the identity of the administered patch. The codes 11 were used for the capsaicin patch, 12 for the control patch and 33 for the lidocaine patch. These codes were retained by a hospital staff member who was not involved in the study and were revealed to the researchers after all the data was collected and analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group LL (Active Comparator): Group LL patients received the 5% lidocaine patch (Lidoderm®, Endo Pharmaceuticals Inc, Malvern, USA) 10 x 14 cm containing 700 mg of Lidocaine for 60 minutes
  Interventions: Drug: Lidocaine 5% patch
- Group LP (Placebo Comparator): Group LP received an identical placebo patch
  Interventions: Drug: Lidocaine 5% patch
- Group LC (Experimental): Group LC received the 8% Capsaicin patch [8% w/w] 640 µg/cm² of adhesive, patch area 280 cm2 (20 cm x 14 cm), (Qutenza®; capsaicin 179 mg patch, Astella Pharma Europe Ltd. Chertsey, UK).
  Interventions: Drug: Capsaicin 8% Patch, Per 10 Square Centimeters

INTERVENTIONS:
Drug: Lidocaine 5% patch — 5% lidocaine patch (Lidoderm®, Endo Pharmaceuticals Inc, Malvern, USA) 10 x 14 cm
  Other Names: Lidocaine patch
  Arms: Group LL; Group LP
Drug: Capsaicin 8% Patch, Per 10 Square Centimeters — 8% Capsaicin patch [8% w/w] 640 µg/cm² of adhesive, patch area 280 cm2 (20 cm x 14 cm), (Qutenza®; capsaicin 179 mg patch, Astella Pharma Europe Ltd. Chertsey, UK)
  Other Names: Capsaicin patch
  Arms: Group LC

SUMMARY:
The study aims to compare the effectiveness and tolerability of using lidocaine 5% patch to 8% capsaicin patch in patients with diabetic neuropathy. Assessment of analgesic effectiveness was assessed by observing any change in the Numeric Pain Rating Scale (NPRS) score, average daily pain Brief Pain Inventory (BPI) for painful diabetic peripheral neuropathy (BPI-DPN Q4) and Patient Global Impression of Change (PGIC). Assessment of capsaicin and lidocaine safety and identifying treatment adverse effects were secondary endpoints in this study

DETAILED DESCRIPTION:
The aim of the present study was to compare the efficacy and tolerability of using lidocaine 5% patch to 8% capsaicin patch in south Asian male patients with diabetic neuropathy. Assessment of analgesic effectiveness was assessed by observing any change in the Numeric Pain Rating Scale (NPRS) score, average daily pain Brief Pain Inventory (BPI) for painful diabetic peripheral neuropathy (BPI-DPN Q4) and Patient Global Impression of Change (PGIC). Assessment of capsaicin and lidocaine safety and identifying treatment adverse effects were secondary endpoints in this study

ELIGIBILITY:
Inclusion Criteria:

* Males aged 40 - 60
* Type 2 diabetes of >10 years duration
* Symptoms of peripheral neuropathic painpresent by scoring on Diabetic neuropathic score (minimum score 1)

Exclusion Criteria:

* Diabetic foot ulcer
* Deformed or contracted foot
* Neurological complications
* Presence of neurological disease
* Presence of cardiovascular or peripheral vascular disease,
* Usage of topical analgesics or implanted medical device six weeks prior to the study

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male only
Enrollment: 290 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Outcome 1 Brief Pain Inventory (BPI) for painful diabetic peripheral neuropathy (BPI-DPN Q4) scores | 24 weeks
  Brief Pain Inventory (BPI) for painful diabetic peripheral neuropathy (BPI-DPN Q4) scores. diabetes at its worst over the past 24 hours").
  Each BPI item uses a 0-10 numeric rating scale anchored at zero for "no pain" and 10 for "pain as bad as you can imagine" for Severity, and "does not interfere" to "completely interferes" for Interference.
Outcome 2 Patient Global Impression of Change score | 24 weeks
  Patient Global Impression of Change score. PGIC is a 7 point scale depicting a patient's rating of overall improvement. The PGIC was patient-reported, and asked the subject to "indicate how you feel now, compared to how you felt before receiving treatment in this study" on a 7-point scale of -3 (very much worse), 0 (no change), to +3 (very much improved).

CONTACTS AND LOCATIONS:
Locations (1):
- Zainab Khan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) can be provided by the author upon reasonable request